CLINICAL TRIAL: NCT07384169
Title: The Impact of Frailty and Different Sedation Techniques on Cognitive Function in Geriatric Colonoscopy Patients
Brief Title: Cognitive Function in Geriatric Colonoscopy Patients
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E2-23-4566
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cognition; Sedation; Geriatric Anesthesia; Frailty; Colonoscopy
Keywords: FRAIL; COGNITIVE FUNCTION; GERIATRIC ANESTHESIA; COLONOSKOPY
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Propofol: Aged 65 years and older who received propofol
  Interventions: Drug: Propofol Group
- Dexmedetomidine: Aged 65 years and older who received dexmedetomidine
  Interventions: Drug: Dexmedetomidine group

INTERVENTIONS:
Drug: Propofol Group — To evaluate cognitive function, Mini Mental State Examination (MMSE) was administered 3 times before the procedure and 2 hours and 24 hours after the procedure. Frailty level of the patient was determined using the frail frailty questionnaire. Each patient received 0.5µg/kg fentanyl (iv).propofol loading dose: 0.2-0.5 mg/kg, continued as repeated boluses for maintenance.
  Other Names: P Group
  Groups: Propofol
Drug: Dexmedetomidine group — To evaluate cognitive function, Mini Mental State Examination (MMSE) was administered 3 times before the procedure and 2 hours and 24 hours after the procedure. Frailty level of the patient was determined using the frail frailty questionnaire. Each patient received 0.5µg/kg fentanyl (iv).The patient was administered a loading dose of dexmedetomidine 0.5 μg/kg-1 over 10 minutes. Propofol 0.1 μg/kg bolus was administered to patients as needed.
  Other Names: D Group
  Groups: Dexmedetomidine

SUMMARY:
Procedures such as colonoscopy cause discomfort and pain and are therefore performed under sedation and analgesia. Although patients aged 65 and older frequently undergo colonoscopy procedures, it is unclear to what extent the anesthetic agents administered for sedation and analgesia in this patient group affect neurocognitive functions. Different sedation methods are used in colonoscopy procedures depending on the anesthesiologist's choice. Propofol is an agent frequently used in general anesthesia or for sedation during endoscopic procedures and, compared to inhaled agents, has more positive effects on postoperative cognitive functions. Dexmedetomidine is an alpha receptor agonist and is preferred due to its positive effects on cognitive functions in elderly patients, its lack of respiratory depression, its ability to provide sedation without impairing cooperation, and its analgesic effects. Although there are studies in the literature on the assessment of neurocognitive function in geriatric patients undergoing surgical procedures, the literature is insufficient in terms of studies addressing cognitive assessment after short-term, outpatient, and less invasive procedures such as colonoscopy. This study aimed to observe patients aged 65 years and older who underwent sedoanalgesia for colonoscopy and to compare the effects on cognitive function by administering the mini mental test before and after the procedure to this patient group.

DETAILED DESCRIPTION:
This study was observational and prospective, and included 164 hospitalized patients aged 65 years and older who received propofol or dexmedetomidine for sedation during colonoscopy. Patients were admitted to the preparation room in the endoscopy unit 30 minutes before the start of colonoscopy. The patients' age, education level (divided into two separate categories: one group with high school education and above, and the other group with less education), Body Mass Index (BMI), American Society of Anesthesiologists (ASA) risk status, and comorbidities were recorded. To assess cognitive function, the Mini Mental State Examination (MMSE) was administered by an investigator who was unaware of which sedation agent would be administered. The patient's degree of frailty was determined using the Frailty Questionnaire. The MMSE was repeated 2 hours after the colonoscopy procedure was completed and at 24 hours. Patients were monitored in the post-anesthesia recovery room using the Modified Aldrete Scoring System. Assessment was performed at 2 hours after the Aldrete Score reached 10 points. Colonoscopy procedures were performed in two separate rooms by two anesthesiologists using two different sedation methods. In our study, patients were observed by anesthesiologists independent of the study in these two rooms. Patients in both groups were started with 3 L/min O2 via a nasal cannula upon entering the room. Patients were monitored for heart rate (HR), systolic arterial blood pressure (SABP), diastolic arterial blood pressure (DABP), mean arterial blood pressure (MAP), and arterial oxygen saturation (SpO2), and baseline measurements of hemodynamic variables were recorded at 5 min, 10 min, and 15 min. Both groups received 0.5 µg/kg fentanyl (IV). In the propofol group (P), the propofol loading dose was 0.2-0.5 mg/kg, and maintenance was continued with repeated boluses. In the dexmedetomidine (D) group, a loading dose of 0.5 μg/kg-1 dexmedetomidine was administered over 10 minutes. When necessary, patients receive propofol 0.1mg/kg push. Ramsey score was maintained at level 3-4 for effective sedation. Colonoscopy procedure duration, total propofol and dexmedetomidine amounts used, and additional atropine and ephedrine administered were recorded. Medications were discontinued upon completion of colonoscopy. Patients were evaluated using the Modified Aldrete Score in the postoperative recovery room and then transferred to the ward. Patients were excluded from the study if complications such as bleeding, perforation, respiratory arrest, or cardiac arrest developed due to the colonoscopy or anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Elective colonoscopy
* ASA physical status I-III
* Provision of written informed consent

Exclusion Criteria:

* Second- or third-degree atrioventricular (AV) block
* A recent history of strokes
* Severe hypotension
* Cardiorespiratory instability
* Substance abuse
* Psychotic illness
* Severe dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 65 years and older
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Assessment of Cognitive Function | Baseline (pre-procedure), 2 hours post-procedure, and 24 hours post-procedure
  Change in cognitive function assessed by Mini Mental State Examination scores. Mini Mental State Examination scores can be between 0-30.
  >10 severe impairment, 10-19 moderate dementia 19-24 early dementia 25 ≤normal

SECONDARY OUTCOMES:
Frailty Score | Baseline (pre-procedure)
  Frailty was assessed using the Clinical Frailty Scale prior to colonoscopy. Frail scores can be between 0-5.
  O normal, 1-2 Pre-frail, 3-5 Frail

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Kaya, M.D., Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share results after published for one year
Supporting Information: CSR
Time Frame: one year
Access Criteria: researchers

REFERENCES:
- [Result] Chen M, Sun Y, Li X, Zhang C, Huang X, Xu Y, Gu C. Effectiveness of single loading dose of dexmedetomidine combined with propofol for deep sedation of endoscopic retrograde cholangiopancreatography (ERCP) in elderly patients: a prospective randomized study. BMC Anesthesiol. 2022 Mar 28;22(1):85. doi: 10.1186/s12871-022-01630-8. PMID 35346041
- [Result] Mei B, Xu G, Han W, Lu X, Liu R, Cheng X, Chen S, Gu E, Liu X, Zhang Y; Perioperative Neurocognitive Disorders (PND) Study Group. The Benefit of Dexmedetomidine on Postoperative Cognitive Function Is Unrelated to the Modulation on Peripheral Inflammation: A Single-center, Prospective, Randomized Study. Clin J Pain. 2020 Feb;36(2):88-95. doi: 10.1097/AJP.0000000000000779. PMID 31714323
- [Result] Qian XL, Zhang W, Liu MZ, Zhou YB, Zhang JM, Han L, Peng YM, Jiang JH, Wang QD. Dexmedetomidine improves early postoperative cognitive dysfunction in aged mice. Eur J Pharmacol. 2015 Jan 5;746:206-12. doi: 10.1016/j.ejphar.2014.11.017. Epub 2014 Nov 20. PMID 25460022
- [Result] Allampati S, Wen S, Liu F, Kupec JT. Recovery of cognitive function after sedation with propofol for outpatient gastrointestinal endoscopy. Saudi J Gastroenterol. 2019 May-Jun;25(3):188-193. doi: 10.4103/sjg.SJG_369_18. PMID 30618439

DOCUMENTS (1):
  • Study Protocol (2023-06-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT07384169/Prot_001.pdf